CLINICAL TRIAL: NCT02187640
Title: A Randomised Controlled Trial of Self-administered Acupressure in Adult Psychiatric Patients With Constipation
Brief Title: Effects of Self-administered Acupressure in Psychiatric Patients With Constipation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Chien Wai-Tong, Professor and Associate Head, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hkpusn01
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Constipation
Keywords: Acupressure; Self-administration; Psychiatric in-patients; Constipation; Self-administered acupressure program; Sham control group
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-administered acupressure (Experimental): A 10-day self-administered acupressure program was implemented by the participants who were adult psychiatric in-patients and randomly assigned into this treatment group. The patients would receive a 3-session training of this therapy conducted by a qualified acupressure therapist and each session lasted about an hour. They would be assessed by the trainer to ensure that they are able to identify the five acupoints and applied a constant and an appropriate pressure on each acupoint before actual implementation.
  Interventions: Behavioral: Self-administered acupressure
- Sham control group (Sham Comparator): Sham control group: Patients would receive 3-session training and be assessed by the trainer. However, they would be trained to locate five non-acupoints adjacent to the actual acupoints and with minimal pressure applied.
  Interventions: Behavioral: Sham control group

INTERVENTIONS:
Behavioral: Self-administered acupressure — Self-administered acupressure: In order to ensure the compliance of treatment, they would apply this intervention according to the acupressure group protocol once per day in groups with one trained research nurse's instructions and supervision .
  Other Names: Self-help acupressure therapy
  Arms: Self-administered acupressure
Behavioral: Sham control group — Sham intervention: Patients received similar aupressure intervention on the non-acupoints.
  Arms: Sham control group

SUMMARY:
This study is to evaluate the effects of self-administered acupressure therapy for psychiatric in-patients with constipation

Two main research questions include:

1. What are the effects of the standardized self-administered acupressure program on reducing those adult psychiatric patients' symptoms of constipation?
2. What are the psychiatric patients' (participants') perceived benefits and limitations of self-administered acupressure on management of their constipation?

In this study, the participants who met the study criteria and completed the baseline measurement would be randomly assigned into either the self-administered acupressure program, or a sham control group who receive a placebo, non-acupoint pressure. The null hypotheses of this study are:

1. There is no significant difference between the acupressure and sham group immediately and/or two weeks after the completion of intervention on patients' symptom severity of constipation; and
2. There is no significant difference between the acupressure and sham group on patients' perceived quality of life at immediately and two weeks after treatment completion.

DETAILED DESCRIPTION:
Main outcomes of this study include the Constipation Assessment Scale (CAS), Patient Assessment Constipation Quality of Life Questionnaire (PAC-QoL), and the socio-demographic and clinical data collected by a trained assessor who was blind to the intervention assignment of the participants. These data would be measured at recruitment (baseline) and immediately (Post-test 1) and two weeks (Post-test 2) after completion of the 10-day intervention. Qualitative focus group interview data would be collected after Post-test 2 .

ELIGIBILITY:
Inclusion criteria of psychiatric in-patients are:

1. Hong Kong Chinese residents, aged 18 to 64 years;
2. satisfied with Rome III diagnostic criteria for constipation; and
3. mentally stable and competent for self-care and learning acupressure, as recommended by their attending psychiatrists.

Exclusion criteria of those in-patients are:

1. anatomical and physiological disorders of gastrointestinal tract such as malrotation, fistula and colonic neuropathies;
2. metabolic and endocrine diseases;
3. lead poisoning and vitamin D intoxication;
4. previous training in acupressure;
5. physical disability involved the upper limbs;
6. planned surgery undergoing during study period; and
7. pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Constipation Assessment Scale | Baseline (0 week; before start of intervention)
  The 8-item Constipation Assessment Scale is an universal measurement tool for symptom severity of constipation in a wide variety of acute and chronic diseases and rated on a 3-point likert scale, ranging from '0= no problem', 1= some problem', and '2= severe problem'. A higher total score will indicate the more severe condition of one's constipation.
Constipation Assessment Scale | Fifth weeks (i.e., immediately after completion of the 10-day intervention)
  The 8-item Constipation Assessment Scale is an universal measurement tool for symptom severity of constipation in a wide variety of acute and chronic diseases and rated on a 3-point likert scale, ranging from '0= no problem', 1= some problem', and '2= severe problem'. A higher total score will indicate the more severe condition of one's constipation.
Constipation Assessment Scale | Seventh week (i.e., two weeks after completion of the intervention)
  The 8-item Constipation Assessment Scale is an universal measurement tool for symptom severity of constipation in a wide variety of acute and chronic diseases and rated on a 3-point likert scale, ranging from '0= no problem', 1= some problem', and '2= severe problem'. A higher total score will indicate the more severe condition of one's constipation.

SECONDARY OUTCOMES:
Patient Assessment Constipation Quality of Life Questionnaire | Baseline (0 week; before start of intervention)
  The Patient Assessment Constipation Quality of Life Questionnaire is a self-administered questionnaire for assessment of the magnitude and degree of interference associated with constipation symptomatology. The scale is composed of 28 items categorized into four subscales, including dissatisfaction (5 items), physical discomfort (4 items), psychosocial discomfort (8 items), and worries and concerns (11 items). Subjects rate each item on a 5-pont likert scale, ranging from '0 = none of the time or not at all to 4 = all of the time or extremely'. The overall and subscale scores can range from 0 to 4, with a lower total score indicating a better health-related quality of life.
Patient Assessment Constipation Quality of Life Questionnaire | Fifth week (i.e., immediately after completion of the 10-day intervention)
  The Patient Assessment Constipation Quality of Life Questionnaire is a self-administered questionnaire for assessment of the magnitude and degree of interference associated with constipation symptomatology. The scale is composed of 28 items categorized into four subscales, including dissatisfaction (5 items), physical discomfort (4 items), psychosocial discomfort (8 items), and worries and concerns (11 items). Subjects rate each item on a 5-pont likert scale, ranging from '0 = none of the time or not at all to 4 = all of the time or extremely'. The overall and subscale scores can range from 0 to 4, with a lower total score indicating a better health-related quality of life.
Patient Assessment Constipation Quality of Life Questionnaire | Seventh week (i.e., two weeks after completion of the 10-day intervention)
  The Patient Assessment Constipation Quality of Life Questionnaire is a self-administered questionnaire for assessment of the magnitude and degree of interference associated with constipation symptomatology. The scale is composed of 28 items categorized into four subscales, including dissatisfaction (5 items), physical discomfort (4 items), psychosocial discomfort (8 items), and worries and concerns (11 items). Subjects rate each item on a 5-pont likert scale, ranging from '0 = none of the time or not at all to 4 = all of the time or extremely'. The overall and subscale scores can range from 0 to 4, with a lower total score indicating a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Kit Wong, MN, DHSc, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- One Regional Mental Hospital, Tuenmen, New Territories, Hong Kong

REFERENCES:
- [Result] 1. Wong, W.K., & Chien, W.T. (2014). Evaluation the effect of Acupressure protocol on Adult psychiatric in-patients with constipation (Program book p. 55). The 35th International Association for Human Caring Conference - 'The Universality of Caring' (24 - 28 May 2014). Kyoto International Conference Center, Kyoto. Division of Family Health Care Nursing, Kobe University Graduate School of Health Sciences, Japan.
- [Derived] Wong WK, Chien WT, Lee WM. Self-administered acupressure for treating adult psychiatric patients with constipation: a randomized controlled trial. Chin Med. 2015 Nov 3;10:32. doi: 10.1186/s13020-015-0064-7. eCollection 2015. PMID 26535053